CLINICAL TRIAL: NCT04596280
Title: Comparision Among Classifications for Acute Diverticulitis: a Multicenter Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Collaborators: San Filippo Neri General Hospital (Other); Hospital San Jacopo (Unknown); Azienda Sanitaria Universitaria Giuliano Isontina (ASU GI) (Unknown)
Responsible Party: Principal Investigator, Dario Tartaglia, Ph.D.; M.D., Researcher, Principal investigator, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: DT - 01- 2020
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Acute Diverticulitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hinchey Classification
  Interventions: Procedure: Colonic Resection
- AAST classification
  Interventions: Procedure: Colonic Resection
- WSES classfication
  Interventions: Procedure: Colonic Resection

INTERVENTIONS:
Procedure: Colonic Resection — Resection of the colonic tract which has been interested by the acute diverticulitis

SUMMARY:
Even though Hinchey classification requires operative intervention, yet remains the established and most universally used scoring system for acute diverticulitis. Several other classifications have been described. The American Association for the Surgery of Trauma (AAST) developed a severity scale for surgical conditions, including diverticulitis. The same was done by the World Society of Emergency Surgery, that proposed a specific classification mainly based on the CT scan findings. This is a pilot study to compare the AAST and WSES classifications for acute colonic diverticulitis with the traditional Hinchey classification. We hypothesize that all the classifications are equivalent one each other in predicting outcomes

ELIGIBILITY:
Inclusion Criteria:

* acute colonic diverticulitis

Exclusion Criteria:

* Other severe conditions of end-life

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Colonic Diverticulitis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Need for procedural intervention (operation or percutaneous drainage) | 30 day

SECONDARY OUTCOMES:
ICU requirement | 30 day
Overall morbidity | 30 day
Length of stay | 30 day
in-hospital morbidity | 30 day

CONTACTS AND LOCATIONS:
Locations (1):
- AOUPisana, Pisa, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: Undecided